CLINICAL TRIAL: NCT05504551
Title: Effect of Superficial Cervical Plexus Block on Incidence and Severity of Post Operative Nausea and Vomiting in Tympanomastoid Operations in Adults, Randomized Controlled Study
Brief Title: Effect of Superficial Cervical Plexus Block on Post Operative Nausea and Vomiting in Tympanomastoid Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wael El-Siory, Lecturer of anesthesia and intensive care medicine- Faculty of Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N-90-2019/MD
Record Dates: First submitted 2022-08-14; First posted 2022-08-17 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: nause, vomiting, tympanomastoid operations
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting

STUDY DESIGN:
Intervention Model Description: study group receives superficial cervical plexus block with lidocaine and bupivacaine control group receives superficial cervical plexus block using normal saline as a placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group B (Active Comparator): Superficial cervical plexus block (SCP) block is given using high frequency linear ultrasound probe connected to an ultrasound machine to visualize superficial cervical plexus (SCP) posterior to the midpoint of sterno cleido mastoid (SCM) muscle. Once SCP is identified, a combination of 5 ml bupivacaine (0.5%) and 5 ml lidocaine (2%) is injected after negative aspiration followed by injection of 1 ml to confirm the area, using a 22 gauge B-bevel Echogenic Needle.
  Interventions: Procedure: ultrasound guided superficial cervical plexus block
- group S (Placebo Comparator): SCP block is given using high frequency linear ultrasound probe connected to an ultrasound machine to visualize SCP posterior to the midpoint of SCM muscle. Once SCP is identified, 10 ml of normal saline is injected after negative aspiration followed by injection of 1 ml to confirm the area, using a 22 gauge B-bevel Echogenic Needle.
  Interventions: Procedure: ultrasound guided superficial cervical plexus block

INTERVENTIONS:
Procedure: ultrasound guided superficial cervical plexus block — SCP block is given using high frequency linear ultrasound probe connected to an ultrasound machine to visualize SCP posterior to the midpoint of SCM muscle. Once SCP is identified, a combination of 5 ml bupivacaine (0.5%) and 5 ml lidocaine (2%) are injected after negative aspiration followed by injection of 1 ml to confirm the area, using a 22 gauge B-bevel needle Echogenic Needle.

SUMMARY:
post operative nausea and vomiting are very common after tympanomastoid operations, in this study we are investigating the effect of superficial cervical plexus block on the incidence and severity of those post operative complications.

DETAILED DESCRIPTION:
various treatments and regimens have been tried to overcome the problem of postoperative nausea and vomiting after tympanomastoid surgery. superficial cervical plexus block seems so promising in this regards as it may reduce the incidence and severity of PONV through 3 mechanisms: primarily through blocking vagal afferents to the middle ear which mediate the vomiting reflex, and secondarily through decreasing pain which aggravates PONV, and finally through decreasing intra and post operative opioid consumption due to adequate analgesia which in turn avoids opioids side effects including PONV.

the study group will receive superficial cervical plexus block while the control will receive the same block while given placebo instead of (lidocain/bupivacaine mixture) incidence and severity of PONV will be recoded according to a scale to find the difference between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients belonging to American Society of Anesthesiologists physical status I-II.
* operation time less than 4 hours.

Exclusion Criteria:

* • American Society of Anesthesiology (ASA) physical status ≥ III.

  * Uncooperative or mentally retarded patients.
  * Known Allergy or hypersensitivity to lidocaine or bupivacaine.
  * Patients known to have gastritis or Gastro-oesophageal reflux disease (GERD).
  * History of PONV or motion sickness.
  * Operation duration (short less than 30 minutes or prolonged more than 240 min).
  * Patients with chronic renal disease (serum creatinine level ≥2.0mg/dl) or on renal replacement therapy (dialysis).
  * Patients with chronic cholecystitis (history of recurrent or persistent vomiting)
  * Skin inflammation and cellulitis.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
PONV incidence over 24hour postoperative | 24 hours
  incidence of PONV according to PONV score from 0 to 3 where: 0= No nausea,no vomiting, 1= Nausea present, no vomiting, 2= Nausea present, vomiting present, 3= Vomiting>2 episodes in 30 minutes, i.e., number of patients with PONV score of 0, number of patients with PONV score of 1, number of patients with PONV score of 2 and number of patients with PONV score of 3.

SECONDARY OUTCOMES:
post operative pain score measured by visual analogue score (VAS) from 0 to 10, where 0= no pain and 10= unbearable pain. | up to 24 hours postoperative
  post operative pain is assessed by visual analogue score from 0 to 10. patients are educated that 0= no pain, 5= distressing pain, 10= unbearable pain.
Intraoperative and postoperative complications | 24 hours
  Complications in the form of bleeding and facial nerve palsy
To monitor intraoperative hemodynamics | up to 4 hours
  To monitor intraoperative heart rate and blood pressure
Side effects and toxicity of drugs | 24 hours
  record any side effects (local anaesthetic lidocaine-bupivacaine) e.g allergy, convulsions, hypotension.
Need for postoperative analgesia | 24 hours
  first analgesic request
To detect complications of regional ear block | 24 hours
  record complications include (hematoma-facial nerve palsy-oedema)

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Elshall, MD, Study Chair — Cairo University
Locations (1):
- Faculty Of Medicine- Cairo Univesity, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apfel CC, Heidrich FM, Jukar-Rao S, Jalota L, Hornuss C, Whelan RP, Zhang K, Cakmakkaya OS. Evidence-based analysis of risk factors for postoperative nausea and vomiting. Br J Anaesth. 2012 Nov;109(5):742-53. doi: 10.1093/bja/aes276. Epub 2012 Oct 3. PMID 23035051
- [Background] Liang S, Irwin MG. Review of anesthesia for middle ear surgery. Anesthesiol Clin. 2010 Sep;28(3):519-28. doi: 10.1016/j.anclin.2010.07.009. Epub 2010 Aug 7. PMID 20850082
- [Background] Cai HD, Lin CZ, Yu CX, Lin XZ. Bilateral superficial cervical plexus block reduces postoperative nausea and vomiting and early postoperative pain after thyroidectomy. J Int Med Res. 2012;40(4):1390-8. doi: 10.1177/147323001204000417. PMID 22971490